CLINICAL TRIAL: NCT04583397
Title: Effects of WiFi Exposure on Sleep and Sleep Related Memory Consolidation in Young Healthy Women
Brief Title: Effects of WiFi Exposure on Sleep in Women
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Corona
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Seibersdorf Labor GmbH (Industry)
Responsible Party: Principal Investigator, Heidi Danker-Hopfe, Head of Competence Center for Sleep Medicine, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EA4/074/19
Record Dates: First submitted 2020-09-24; First posted 2020-10-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: WiFi - Sham (Experimental): first intervention WiFi, second intervention sham
  Interventions: Other: radio frequency electromagnetic fields
- Experimental: Sham - WiFi (Experimental): first Intervention sham, second Intervention WiFi
  Interventions: Other: radio frequency electromagnetic fields

INTERVENTIONS:
Other: radio frequency electromagnetic fields — Exposure system delivers emissions comparable to those from a WiFi access Point close to the bed or sham (no exposure)

SUMMARY:
Effects of Wifi exposure on sleep and sleep-related memory consolidation are investigated in a double-blind, sham-controlled fully counterbalanced study design in young healthy women.

DETAILED DESCRIPTION:
Introduction: Since several years Wireless Local Networks (WLAN, WiFi) are widely spread and operated in households. Many people feel that the presence of radiofrequency technologies impairs their health. Sleep problems are among the most often complained complaints. The present study aims to contribute to answer the question, whether biological effects of a WiFi exposure can be assessed by objective measures. The results of this study will expand the database on possible acute effects of WiFi exposure and thus qualitatively contribute to the discussion whether sleep is affected by exposure from radiofrequency electromagnetic fields.

Methods: A double-blind, sham-controlled experiment in the sleep laboratory with exposure conditions delivered in a balanced randomized cross-over design. Subjective sleep quality of volunteers is assessed by questionnaires. Macro- and microstructure of sleep are measured by polysomnography. Furthermore, a possible impact on sleep related memory consolidation is tested. To do so declarative, procedural and emotional memory tasks are used. Exposure is delivered by a specially developed system, which simulates field strengths and signals occurring in a subject sleeping in the close proximity of a WiFi-access point. This exposure system is necessary to allow for a double-blind implementation and monitoring as well as for the realization of defined exposure parameters.

The study aims to analyse possible sex differences in WiFi exposure effects on sleep and sleep related memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Only right-handed
* non-smokers
* Pittsburgh Sleep Quality Index (PSQI) score < 5
* no extreme morning/evening preference [Morningness-Eveningness Questionnaire (MEQ) score ≥ 31 or ≤ 69
* no indication of depression or somatic symptoms as assessed by a medical examination and validated questionnaires [Patient Health Questionnaires (PHQ-9 and PHQ-15) scores ≤ 5 and ≤ 10, respectively

Exclusion Criteria:

* history of a psychiatric disorder,
* history of a neurological and/or sleep disorder
* excessive daytime sleepiness [Epworth Sleepiness Scale (ESS) score > 9;
* non-regular sleep-wake schedule as assessed by a sleep diary
* a regular intake of medication that affects the central nervous system, excessive caffeine and/or alcohol consumption, regular and occasional drug use,
* metal implants
* periodic leg movement arousal index > 10/h in the Adaptation night
* apnoea-hypopnoea-index > 5/h in the Adaptation night.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only women will be included, a corresponding study for men has already been completed
Enrollment: 34 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency index | 8 hours
  (total Sleep time in % of time in bed)

SECONDARY OUTCOMES:
declarative memory | 8 hours
  number of remembered word pairs in the Word Association Task
Sleep EEG power | 8 hours
  EEG power in the spindle frequency range

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No